CLINICAL TRIAL: NCT00263354
Title: Oxaliplatin Phase II Trial in Association With 5FU and Folinic Acid in the Treatment of Advanced Unresectable or Metastatic Gastric Cancer.
Brief Title: Oxaliplatin in Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8915
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-08

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin

SUMMARY:
To determine the objective response to oxaliplatin/5FU/leucovorin combination chemotherapy in patients with advanced unresectable or metastatic gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0-2.
* Histologically proven gastric or gastro-esophageal junction adenocarcinoma.
* At least unidimensional measurable disease. If a unique metastasis constitutes the only disease sign, it requires histological confirmation.
* First line locally unresectable or metastatic gastric cancer.
* Relapsing gastric cancer after local and/or systemic treatment with a post-surgical period of at least 4 weeks, a post-adjuvant or neoadjuvant chemoradiotherapy period of at least 6 months.
* Serum bilirubin < 2 mg/dl
* Serum creatinine < or = 2 mg/dl
* Hemoglobin > or = 10 g/dl
* Absolute neutrophil count > or = 2000/dl
* Platelet count >or = 100, 000/dl
* AST/ALT < or = 2.5 time-fold the institutional normal upper limit
* Alkaline phosphatase < or = 5 time-fold the institutional normal upper limit
* Imagenological evaluation of the patient at least 2 weeks prior to the drug infusion
* Laboratory tests at least 1 week prior to the first infusion
* Patient available for follow up and able to answer to the quality of life questionnaire

Exclusion Criteria:

* Symptomatic sensorial peripheral neuropathy
* Uncontrolled concomitant disease
* Another malignant neoplastic disease diagnosed within the previous 5 years to the diagnosis of advanced or metastatic gastric cancer, with the exception of 'in situ' cervix carcinoma or non-melanoma skin cancer
* Concomitant antitumoral treatment
* Cerebral metastases
* Unstable heart disease, even though in treatment
* Myocardial infarction within the last 6 months
* Radiotherapy within the last 6 weeks, surgery within the last 4 weeks, or chemotherapy within the last 6 months.
* Pregnancy or nursing ( or women in reproductive life without adequate contraception)
* Significant neurological or psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To evaluate response rate according to RECIST criteria
To evaluate the progression-free survival in the ITT population

SECONDARY OUTCOMES:
To evaluate the overall survival in the ITT population
To investigate safety using NCI-CTC criteria version 2

CONTACTS AND LOCATIONS:
Overall Officials: Jesus M. Ruiz, MD, Study Director — Sanofi